CLINICAL TRIAL: NCT04498936
Title: Efficacy of Adding Sofosbuvir/Ledipasvir Combination, or Nitazoxanide to the Standard of Care in Treatment of COVID-19: A Randomized Controlled Trial
Brief Title: Sofosbuvir/Ledipasvir and Nitazoxanide for Treatment of COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Helwan University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Medhat, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19 treatment
Record Dates: First submitted 2020-04-14; First posted 2020-08-05 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: COVID
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination; Therapeutics; nitazoxanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sofosbuvir/Ledipasvir (Experimental): This group will receive a fixed combination of Sofosbuvir/Ledipasvir (400 mg and 90 mg, orally) once daily for 14 days, plus the standard care treatment regimen (SCT) for COVID-19 patients according to the Egyptian Ministry of Health (MOH) protocol.
  Interventions: Drug: Sofosbuvir and Ledipasvir
- Nitazoxanide (Experimental): This group will receive nitazoxanide (500 mg, orally) four times per day for 14 days, plus the standard care treatment regimen (SCT) for COVID-19 patients according to the Egyptian Ministry of Health (MOH) protocol.
  Interventions: Drug: Nitazoxanide
- Standard care treatment (No Intervention): This group will receive only the standard care treatment regimen (SCT) for COVID-19 patients according to the Egyptian Ministry of Health (MOH) protocol.

INTERVENTIONS:
Drug: Sofosbuvir and Ledipasvir — Evaluate the efficacy of Sofosbuvir/Ledipasvir in treatment of COVID-19
  Other Names: Treatment
  Arms: Sofosbuvir/Ledipasvir
Drug: Nitazoxanide — Evaluate the efficacy of Nitazoxanide in treatment of COVID-19
  Other Names: Treatment
  Arms: Nitazoxanide

SUMMARY:
The efficacy of treating COVID-19 infection by using Sofosbuvir/Ledipasvir and Nitazoxanide will be examined. Included patients will be into 3 groups. The 1st group will receive Sofosbuvir/Ledipasvir plus the standard care treatment (SCT). The 2nd group will take Nitazoxanide and SCT, while the 3rd group will receive only SCT. Then the clinical improvement and the rate of PCR change from positive to negative will be evaluated in each group.

DETAILED DESCRIPTION:
This study is an open-label, randomized, controlled trial. A total of 240 patients who are recruited in 2 quarantine hospitals (15th of May hospital, Cairo, and Al Rajhi hospital, Assiut), will be randomly assigned in a 1:1:1 ratio (80 patient in each treatment arm), to receive either the fixed combination of Sofosbuvir/Ledipasvir (400 mg and 90 mg, orally) once daily for 14 days, plus the standard care treatment regimen (SCT) for COVID-19 patients according to the Egyptian Ministry of Health (MOH) protocol (Group 1), or nitazoxanide (500 mg, orally) four times per day for 14 days, plus STC (Group 2), or SCT alone (Group 3). All treatment groups will be followed up by laboratory investigations and PCR for SARS-CoV-2 virus at the time of enrollment, days 5, 8, 11, and 14. Supportive care comprised, as necessary, supplemental oxygen, noninvasive and invasive ventilation, antibiotic agents, vasopressor support, renal-replacement therapy, and extracorporeal membrane oxygenation (ECMO). To ensure a balanced distribution of case severities in all study groups, randomization will be stratified based on the case severity index issued by WHO (https://www.who.int/docs/default-source/coronaviruse/clinical-management-of-novel-cov.pdf).

Written informed consent will be obtained from all patients or the patient's legal representative if the patient is too unwell to provide consent. The trial will be conducted in accordance with the principles of the Declaration of Helsinki and the Good Clinical Practice guidelines of the International Conference on Harmonisation. The authors are responsible for designing the trial and for compiling and analyzing the data. The authors vouch for data completeness and accuracy and adherence to the trial protocol.

ELIGIBILITY:
This study is an open-label, randomized, controlled trial. A total of 216 patients who are recruited in 2 quarantine hospitals (15th of May hospital, Cairo, and Al Rajhi hospital, Assiut), will be randomly assigned in a 1:1:1 ratio (72 patient in each treatment arm), to receive either the fixed combination of Sofosbuvir/Ledipasvir (400 mg and 90 mg, orally) once daily for 14 days, plus the standard care treatment regimen (SCT) for COVID-19 patients according to the Egyptian Ministry of Health (MOH) protocol (Group 1), or nitazoxanide (500 mg, orally) four times per day for 14 days, plus STC (Group 2), or SCT alone (Group 3). All treatment groups will be followed up by laboratory investigations and PCR for SARS-CoV-2 virus at the time of enrollment, days 5, 8, 11, and 14. Supportive care comprised, as necessary, supplemental oxygen, noninvasive and invasive ventilation, antibiotic agents, vasopressor support, renal-replacement therapy, and extracorporeal membrane oxygenation (ECMO). To ensure a balanced distribution of case severities in all study groups, randomization will be stratified based on the case severity index issued by WHO (https://www.who.int/docs/default-source/coronaviruse/clinical-management-of-novel-cov.pdf).

Written informed consent will be obtained from all patients or the patient's legal representative if the patient is too unwell to provide consent. The trial will be conducted in accordance with the principles of the Declaration of Helsinki and the Good Clinical Practice guidelines of the International Conference on Harmonisation. The authors are responsible for designing the trial and for compiling and analyzing the data. The authors vouch for data completeness and accuracy and adherence to the trial protocol.

Inclusion Criteria:

* This study will include patients with confirmed COVID-19 infection and admitted to COVID-19 quarantine hospitals. Included patients should be > 12 years old, with creatinine clearance > 30 mL/ml, and without any malignancy. Patients with COVID-19 infection are classified clinically into mild, moderate, severe, and critical cases according to the management guide for COVID-19 published by the Egyptian Ministry of Health and Population. Mild cases are defined as patients in whom clinical symptoms are mild, and no pneumonia manifestations can be found in imaging. Moderate cases are defined as patients having symptoms such as fever and respiratory tract symptoms, etc. and pneumonia manifestations can be seen in imaging. Severe cases are patients who meet any of the following criteria; (a) respiratory rate > 30 breaths/min, (b) oxygen saturations< 93% at a rest state, (c) arterial partial pressure of oxygen (PaO2)/ Fraction of inspired oxygen (FiO2)<300 mm Hg, or (d) patients with more than 50% lesions progression within 24 to 48 hours in lung imaging should be treated as severe cases. Finally, critical patients are those who are meeting any of the following criteria; (a) occurrence of respiratory failure requiring mechanical ventilation, or (b) the presence of shock; other organ failures that require monitoring and treatment in the ICU. All patients with an established diagnosis of COVID-19 in Egyptian quarantine hospitals at any clinical stage will be included in this study.

Exclusion Criteria:

* Patients < 12 years old.
* Pregnant females.
* Patients with renal impairment with creatinine clearance < 30 mL/min.
* Patients with malignancies particularly Hepatocellular Carcinoma (HCC).
* Patients using Favipiravir or Lopinavir-Ritonavir, as the co-administration of these drugs with Sofosbuvir/Ledipasvir has not been studied.
* Patients with decompensated liver cirrhosis (Child-Pugh score B and C).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change of PCR from positive to negative | 2 weeks
  The PCR will be done at time of recruitment, day 5, 8, 11, and 14. The time taken to have negative will be measured in each group.
Clinical improvement | 2 weeks
  Clinical improvement will be measured by detection of downgrading of cases severity according to the World Health Organization case severity classification.

SECONDARY OUTCOMES:
Adverse events | 2 weeks
  All patients will be asked about any possible adverse effects that they may suffer from taken drugs during their follow up. Any mentioned side effect will be reported. Drug discontinuation and it cause will be also reported if it happened.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Medhat, PhD, Principal Investigator — Assiut University; Mohamed El Kassas, PhD, Study Chair — Helwan University; Haidi K Ramadan, PhD, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - 15th May Hospital, Helwan, Cairo Governorate
  - Assiut University Hospital, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ju, J., et al., Nucleotide Analogues as Inhibitors of Viral Polymerases. bioRxiv, 2020: p. 2020.01.30.927574.
- [Background] Zumla A, Chan JF, Azhar EI, Hui DS, Yuen KY. Coronaviruses - drug discovery and therapeutic options. Nat Rev Drug Discov. 2016 May;15(5):327-47. doi: 10.1038/nrd.2015.37. Epub 2016 Feb 12. PMID 26868298
- [Background] Elfiky AA. Ribavirin, Remdesivir, Sofosbuvir, Galidesivir, and Tenofovir against SARS-CoV-2 RNA dependent RNA polymerase (RdRp): A molecular docking study. Life Sci. 2020 Jul 15;253:117592. doi: 10.1016/j.lfs.2020.117592. Epub 2020 Mar 25. PMID 32222463
- [Background] Chen YW, Yiu CB, Wong KY. Prediction of the SARS-CoV-2 (2019-nCoV) 3C-like protease (3CL pro) structure: virtual screening reveals velpatasvir, ledipasvir, and other drug repurposing candidates. F1000Res. 2020 Feb 21;9:129. doi: 10.12688/f1000research.22457.2. eCollection 2020. PMID 32194944
- [Background] Mo Y, Fisher D. A review of treatment modalities for Middle East Respiratory Syndrome. J Antimicrob Chemother. 2016 Dec;71(12):3340-3350. doi: 10.1093/jac/dkw338. Epub 2016 Sep 1. PMID 27585965
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] European Association for the Study of the Liver. EASL Recommendations on Treatment of Hepatitis C 2018. J Hepatol. 2018 Aug;69(2):461-511. doi: 10.1016/j.jhep.2018.03.026. Epub 2018 Apr 9. No abstract available. PMID 29650333
- [Background] Wu A, Peng Y, Huang B, Ding X, Wang X, Niu P, Meng J, Zhu Z, Zhang Z, Wang J, Sheng J, Quan L, Xia Z, Tan W, Cheng G, Jiang T. Genome Composition and Divergence of the Novel Coronavirus (2019-nCoV) Originating in China. Cell Host Microbe. 2020 Mar 11;27(3):325-328. doi: 10.1016/j.chom.2020.02.001. Epub 2020 Feb 7. PMID 32035028
- [Background] Frieman M, Baric R. Mechanisms of severe acute respiratory syndrome pathogenesis and innate immunomodulation. Microbiol Mol Biol Rev. 2008 Dec;72(4):672-85, Table of Contents. doi: 10.1128/MMBR.00015-08. PMID 19052324
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Background] Lam KK, Zheng X, Forestieri R, Balgi AD, Nodwell M, Vollett S, Anderson HJ, Andersen RJ, Av-Gay Y, Roberge M. Nitazoxanide stimulates autophagy and inhibits mTORC1 signaling and intracellular proliferation of Mycobacterium tuberculosis. PLoS Pathog. 2012;8(5):e1002691. doi: 10.1371/journal.ppat.1002691. Epub 2012 May 10. PMID 22589723
- [Background] Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. J Infect Public Health. 2016 May-Jun;9(3):227-30. doi: 10.1016/j.jiph.2016.04.001. Epub 2016 Apr 16. PMID 27095301
- [Background] Rossignol JF, La Frazia S, Chiappa L, Ciucci A, Santoro MG. Thiazolides, a new class of anti-influenza molecules targeting viral hemagglutinin at the post-translational level. J Biol Chem. 2009 Oct 23;284(43):29798-808. doi: 10.1074/jbc.M109.029470. Epub 2009 Jul 28. PMID 19638339
- [Background] Cao J, Forrest JC, Zhang X. A screen of the NIH Clinical Collection small molecule library identifies potential anti-coronavirus drugs. Antiviral Res. 2015 Feb;114:1-10. doi: 10.1016/j.antiviral.2014.11.010. Epub 2014 Nov 28. PMID 25451075
- [Background] Padmanabhan, S., Potential dual therapeutic approach against SARS-CoV-2/COVID-19 with Nitazoxanide and Hydroxychloroquine. 2020.
- [Background] Ueda Y, Ikegami T, Akamatsu N, Soyama A, Shinoda M, Goto R, Okajima H, Yoshizumi T, Taketomi A, Kitagawa Y, Eguchi S, Kokudo N, Uemoto S, Maehara Y. Treatment with sofosbuvir and ledipasvir without ribavirin for 12 weeks is highly effective for recurrent hepatitis C virus genotype 1b infection after living donor liver transplantation: a Japanese multicenter experience. J Gastroenterol. 2017 Aug;52(8):986-991. doi: 10.1007/s00535-017-1310-9. Epub 2017 Jan 30. PMID 28138756
- [Background] Liu CJ, Chuang WL, Sheen IS, Wang HY, Chen CY, Tseng KC, Chang TT, Massetto B, Yang JC, Yun C, Knox SJ, Osinusi A, Camus G, Jiang D, Brainard DM, McHutchison JG, Hu TH, Hsu YC, Lo GH, Chu CJ, Chen JJ, Peng CY, Chien RN, Chen PJ. Efficacy of Ledipasvir and Sofosbuvir Treatment of HCV Infection in Patients Coinfected With HBV. Gastroenterology. 2018 Mar;154(4):989-997. doi: 10.1053/j.gastro.2017.11.011. Epub 2017 Nov 22. PMID 29174546
- [Background] Lim YS, Ahn SH, Lee KS, Paik SW, Lee YJ, Jeong SH, Kim JH, Yoon SK, Yim HJ, Tak WY, Han SY, Yang JC, Mo H, Garrison KL, Gao B, Knox SJ, Pang PS, Kim YJ, Byun KS, Kim YS, Heo J, Han KH. A phase IIIb study of ledipasvir/sofosbuvir fixed-dose combination tablet in treatment-naive and treatment-experienced Korean patients chronically infected with genotype 1 hepatitis C virus. Hepatol Int. 2016 Nov;10(6):947-955. doi: 10.1007/s12072-016-9726-5. Epub 2016 May 20. PMID 27198664
- [Background] Fox LM, Saravolatz LD. Nitazoxanide: a new thiazolide antiparasitic agent. Clin Infect Dis. 2005 Apr 15;40(8):1173-80. doi: 10.1086/428839. Epub 2005 Mar 14. PMID 15791519
- [Background] Stockis A, Deroubaix X, Lins R, Jeanbaptiste B, Calderon P, Rossignol JF. Pharmacokinetics of nitazoxanide after single oral dose administration in 6 healthy volunteers. Int J Clin Pharmacol Ther. 1996 Aug;34(8):349-51. PMID 8864798
- See also: Epidemiological data about Covid-19 — https://google.com/covid19-map/?hl=en